CLINICAL TRIAL: NCT05935852
Title: Contrast-enhanced Multispectral Optoacoustic Tomography for Non-invasive Assessment of Diabetic Gastroparesis
Acronym: TRANSPARENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Ferdinand Knieling, PD Dr. med. Ferdinand Knieling, University of Erlangen-Nürnberg Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-TEMP915246-Bm
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Diabetic Gastroparesis
Keywords: diabetic gastroparesis; MSOT

STUDY DESIGN:
Intervention Model Description: Four Arms with different disease activity and duration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study group 1 (Other): Multispectral Optoacoustic Tomography (MSOT) of the gastric antrum and terminal ileum in patients with T1DM, aged> 18 years, with diabetic neuropathy
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)
- Study group 2 (Other): Multispectral Optoacoustic Tomography (MSOT) of the gastric antrum and terminal ileum in patients with T1DM, aged> 18 years, without diabetic neuropathy
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)
- Study group 3 (Other): Multispectral Optoacoustic Tomography (MSOT) of the gastric antrum and terminal ileum in patients with T1DM, aged < 18 years, disease activity 5 - 10 years, HbA1c > 8,5%
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)
- Study group 4 (Other): Multispectral Optoacoustic Tomography (MSOT) of the gastric antrum and terminal ileum in patients with T1DM, aged < 18 years, disease activity 5 - 10 years, HbA1c < 7,5%
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)

INTERVENTIONS:
Device: Multispectral Optoacoustic Tomography (MSOT) — Non-invasive transcutaneous imaging of endogenous and exogenous chromophores via infrared and near-infrared laser pulses

SUMMARY:
The objective of the proposed study is to assess gastric emptying time (GET) based on contrast-enhanced multispectral optoacoustic imaging (CE-MSOT) in a collective of patients with type 1 diabetes mellitus (T1DM). The results will be correlated with disease duration and severity.

DETAILED DESCRIPTION:
T1DM is a chronic autoimmune disease in which autoantibodies destroy the pancreas's insulin-producing cells. In Germany, it is estimated that 32,000 children and adolescents and approximately 335,000 adults suffer from T1DM. The trend has been increasing in recent years.

A complication of T1DM is diabetic gastroparesis (DGP), in which gastric emptying is delayed without mechanical obstruction. Symptoms of DGP include nausea, vomiting, and abdominal pain. Many patients* are asymptomatic.

DGP is associated with higher HbA1c, autonomic neuropathy, nephropathy, retinopathy, and increased gastrointestinal symptoms.

In this study, gastric emptying will be imaged noninvasively and without radiation based on MSOT. MSOT, in addition to imaging endogenous chromophores, allows visualization of exogenous chromophores. If the dye indocyanine green (ICG) is ingested orally, the signal of the dye in the lumen of the gastrointestinal tract can be visualized noninvasively by MSOT over different intestinal segments. If food is labeled with ICG and ingested by subjects*, the passage of chyme through the gastrointestinal tract can be tracked by measuring the signal with MSOT, and transit times can be measured.

This study will investigate gastric emptying times of patients* with T1DM.

ELIGIBILITY:
nclusion criteria Group 1

* Written informed consent
* T1DM diagnosis
* Duration of disease at least 5, preferably 10 years with diagnosed neuropathy Group 2
* Written informed consent
* T1DM diagnosis
* Duration of disease at least 5, preferably 10 years without diagnosed neuropathy Group 3
* Written informed consent from parent or guardian
* T1DM diagnosis
* Duration of disease at least 5, preferably 10 years with inadequate medication control (HbA1c value > 8.5 mmol/l) Group 4
* Written informed consent of parent or guardian
* T1DM diagnosis
* Duration of disease at least 5, preferably 10 years with good medication control (HbA1c value < 7.5 mmol/l) Exclusion criteria

Generality:

* Pregnancy
* Breastfeeding mothers
* Tattoo in the area of the examination
* Subcutaneous fat tissue over 3 cm
* Known hypersensitivity to ICG, sodium iodide or iodine
* Hyperthyroidism, focal or diffuse thyroid autonomy
* Timely close treatment to check thyroid function with ingestion of radioactive iodine (within two weeks before or after the study)
* Impaired renal function
* Taking the following medications: Beta blockers, anticonvulsants, cyclopropane, bisulfite compounds, haloperidol, heroin, meperidine, metamizole, methadone, morphine, nitrofurantoin, opium alkaloids, phenobarbital, phenylbutazone, probenecid, rifamycin, any injection containing sodium bisulfite

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-24 (Estimated)

PRIMARY OUTCOMES:
Gastric emptying time | 6 hours
  Gastric emptying time based on MSOT imaging of ICG-signal intensity

SECONDARY OUTCOMES:
Correlation of acquired hemoglobin signal with disease activity | 6 hours
  Hemoglobin-associated parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT correlated with disease activity
Correlation of acquired hemoglobin signal with disease duration | 6 hours
  Hemoglobin-associated parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT correlated with disease duration

IPD SHARING:
Plan to Share IPD: Undecided